CLINICAL TRIAL: NCT06641531
Title: Prevalence of Abnormal Pap Smear in Sohag University Hospital Outpatient Clinic
Brief Title: Prevalence of Abnormal Pap Smear
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Ahmed Elsayed Radwan, Resident at Obstetrics and Gynecology department Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-24-09-13MS
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal group: normal pap smear
  Interventions: Other: Screening pap smear test
- Abnormal group: Abnormal routine Pap smears will be classified according to latest Bethesda system into the following categories : Atypical squamous cells of undetermined significance (ASC-US), atypical squamous cells cannot exclude high grade squamous intraepithelial lesion (ASC-H), low grade squamous intraepithelial lesion (LSIL), high grade squamous intraepithelial lesion (HSIL), squamous cell carcinoma (SCC), atypical glandular cells of undetermined significance (AGUS), and adenocarcinoma (ADC).
  Interventions: Other: Screening pap smear test

INTERVENTIONS:
Other: Screening pap smear test — The patient put in dorsal lithotomy position and place the feet in stirrups or on foot rests . then, the physician will insert a cusco speculum into the vagina to hold vaginal wall open . The specimens will be collected as follows; firstly, the speculum will be inserted without lubricant. Any mucous, discharge or blood will be removed with dry cotton. A wooden spatula will be used for sampling ectocervix which will be rotated 360 degrees. For sampling endocervix, A brush or a swab will be rotated only 90 degrees as the circumferential bristles will be in contact with the entire surface the moment the brush is inserted.
  The samples will be applied to the slides which will be encoded and immediately fixed in 95% ethanol and the samples will be transferred to pathology department to be stained by the standard Papanicolaou stain

SUMMARY:
This study aims to evaluate prevalence of abnormal Pap smear among sexually active women of reproductive age attending sohag university hospital outpatient clinic.

DETAILED DESCRIPTION:
This study aims to evaluate prevalence of abnormal Pap smear among sexually active women of reproductive age attending Sohag university hospital outpatient clinic. Participating women will be subjected to accurate history taking regarding age, parity, Body mass index, contraceptive use, menstrual history, and duration of marital life, frequency of previous marriages if any, and the status of cervix by per-vaginal examination of the patients.

The patient put in dorsal lithotomy position and place the feet in stirrups or on foot rests . then, the physician will insert a cusco speculum into the vagina to hold vaginal wall open . The specimens will be collected as follows; firstly, the speculum will be inserted without lubricant. Any mucous, discharge or blood will be removed with dry cotton. A wooden spatula will be used for sampling ectocervix which will be rotated 360 degrees. For sampling endocervix, A brush or a swab will be rotated only 90 degrees as the circumferential bristles will be in contact with the entire surface the moment the brush is inserted.

The samples will be applied to the slides which will be encoded and immediately fixed in 95% ethanol and the samples will be transferred to pathology department to be stained by the standard Papanicolaou stain . The Bethesda System will be used for cytological interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant sexually active women aged from 21 to 60 years old.
* Patients who didn't have their pap smear done in last 3 years .
* Patient who had previous abnormal pap smear and coming for follow up.

Exclusion Criteria:

* Women who were diagnosed cervical cancer that was treated.
* Women who underwent total hysterectomy.
* Women who are pregnant.
* Patients whose pap smear was done in last 3 years with reassuring results.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — sexually active women of reproductive age.
Study Population: Non pregnant sexually active women aged from 21 to 60 years old.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
number of abnormal pap smear among sexually active women of reproductive age attending sohag university hospital outpatient clinic. | From October 2024 to April 2025
  to evaluate prevalence of abnormal Pap smear among sexually active women of reproductive age attending sohag university hospital outpatient clinic.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No